CLINICAL TRIAL: NCT02685488
Title: A Pilot Study: Investigating Transcranial Ultrasound as a Potential Intervention for Mild to Moderate Depression
Brief Title: Investigating Transcranial Ultrasound as a Potential Intervention for Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, John Allen, Distinguished Professor, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RSRCH---703FY'15
Record Dates: First submitted 2016-02-14; First posted 2016-02-18 (Estimated); Results first posted 2018-01-08 (Actual); Last update posted 2018-01-08 (Actual); Status verified 2018-01

CONDITIONS: Depression; Anxiety Disorders
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transcranial Ultrasound Power (Active Comparator): Transcranial Ultrasound Power
  Interventions: Device: Transcranial Ultrasound Power
- Transcranial Ultrasound Sham (Sham Comparator): Transcranial Ultrasound Sham. Unknown to both participants and experimenters, the ultrasound will not stimulate.
  Interventions: Device: Transcranial Ultrasound Sham

INTERVENTIONS:
Device: Transcranial Ultrasound Power — Transcranial ultrasound will be to stimulate at the right fronto-temporal cortex. 30 seconds of stimulation at 500 kHZ with duty cycle 0.24% and pulse rate frequency at 40 Hz.
  Arms: Transcranial Ultrasound Power
Device: Transcranial Ultrasound Sham — Transcranial ultrasound will be used without power for a "sham" condition.
  Arms: Transcranial Ultrasound Sham

SUMMARY:
Depression is the leading cause of disability worldwide. Because a significant number of people with depression do not respond to medication or therapy, alternative treatment options are greatly needed. Recent research has focused on brain stimulation methods due to their therapeutic utility for treating depression. Yet, current brain stimulation methods have drawbacks, including invasive surgery and limited precision in targeting specific areas. A novel brain stimulation method, transcranial ultrasound (TUS), is noninvasive, has greater spatial precision than most existing methods, and is proven safe for humans. TUS has been found to increase positive mood in chronic pain patients. In a double blind study, TUS increased positive mood in over 140 healthy undergraduates at the University of Arizona.

Despite evidence that TUS can increase positive mood in humans, it has yet to be investigated whether TUS can increase positive mood in humans who are experiencing chronic low mood or depression. The present study will, for the first time, examine whether TUS can improve depressive symptoms. Twenty to thirty participants with mild to moderate depressive symptoms (Beck Depression Inventory Score between 10 and 25) will be randomly assigned to a TUS sham or TUS activation condition. In the TUS activation condition, TUS will be used to stimulate the right fronto-temporal area, which has previously been shown to increase positive mood. Participants in the TUS sham condition will not receive any brain stimulation. Participants will attend five sessions within seven days or ten sessions within fourteen days. At each session, in addition to brain stimulation, self-reported mood and depressive symptoms will be recorded. Furthermore, the investigators will use electroencephalogram (EEG) to record changes in brain electrical signals during TUS stimulation. Based on prior research, the investigators predict that mood will increase and depressive symptoms will decrease with TUS stimulation.

DETAILED DESCRIPTION:
Participants will first complete the online screening and those who qualify to complete the study will be contacted via telephone (see above for telephone recruitment and consent procedure). After providing informed consent, on the first day, participants will be randomly assigned to either a TUS treatment or a TUS sham condition (placebo), and the study will be double blind. Participants in the TUS treatment condition (with sham or treatment unknown to both participant and experimenter) will have TUS stimulation at the right fronto-temporal area five times within seven days or ten times within fourteen days.

Participants will sign up for the first five sessions first but will be reminded participants may withdraw from the study at any time. Should participants choose to continue with the second week of treatment, participants will be scheduled for another five sessions. In other words, participants will have the option of completing 10 days of the procedure. The procedure does not differ between week 1 and week 2. However, participants will be compensated less for week 2. Participants will have the option to continue into week 2, as participants may find that the treatment is benefiting them. The first, fifth, and tenth days of the study will take approximately 2 hours and the second, third, fourth, sixth, seventh, eighth, and ninth will take only one hour.

In the sham condition, the ultrasound probe will be placed at the right fronto-temporal area five times over the course of seven days or ten times over the course of fourteen days without the stimulation. Prior research has shown that stimulation at this area induces positive mood change and is implicated in positive mood. On the first, middle, and last day of the procedure (day 1, 5, 10), EEG data will be collected. On the second, third, and fourth day as well as sixth through ninth days of the procedure EEG data will not be collected and only TUS stimulation will occur. Collecting EEG data at these points will allow for comparison of resting electrical brain profiles from the beginning of the study to the end of the study. Additionally, the investigators will assess state mood and rumination before and after TUS, as well as depressive and anxiety symptoms at the end of each day. The state mood and rumination will allow us to examine the mood effects of TUS, whereas the depressive and anxiety symptoms questionnaires will allow us to examine any changes in these important profiles over the course of the study.

ELIGIBILITY:
Inclusion Criteria:

* Beck Depression Inventory score between 10 and 25

Exclusion Criteria:

* left-handedness
* prior serious head-related injury
* any medical condition that would impact EEG profiles
* chronic migraines or other severe headaches
* pregnancy
* lack of proficiency in English
* lack of secure housing
* current confounding treatment (including any psychotropic medication or psychotherapy)
* current active suicidal potential necessitating immediate treatment, as such participants will be referred for immediate treatment.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2015-10; Primary Completion 2016-04 (Actual); Study Completion 2016-05 (Actual)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hameroff S, Trakas M, Duffield C, Annabi E, Gerace MB, Boyle P, Lucas A, Amos Q, Buadu A, Badal JJ. Transcranial ultrasound (TUS) effects on mental states: a pilot study. Brain Stimul. 2013 May;6(3):409-15. doi: 10.1016/j.brs.2012.05.002. Epub 2012 May 29. PMID 22664271
- [Background] Tufail Y, Yoshihiro A, Pati S, Li MM, Tyler WJ. Ultrasonic neuromodulation by brain stimulation with transcranial ultrasound. Nat Protoc. 2011 Sep 1;6(9):1453-70. doi: 10.1038/nprot.2011.371. PMID 21886108
- [Background] Fava M. Diagnosis and definition of treatment-resistant depression. Biol Psychiatry. 2003 Apr 15;53(8):649-59. doi: 10.1016/s0006-3223(03)00231-2. PMID 12706951
- [Background] Gavrilov LR, Tsirulnikov EM, Davies IA. Application of focused ultrasound for the stimulation of neural structures. Ultrasound Med Biol. 1996;22(2):179-92. doi: 10.1016/0301-5629(96)83782-3. PMID 8735528
- [Background] Bystritsky A, Korb AS, Douglas PK, Cohen MS, Melega WP, Mulgaonkar AP, DeSalles A, Min BK, Yoo SS. A review of low-intensity focused ultrasound pulsation. Brain Stimul. 2011 Jul;4(3):125-36. doi: 10.1016/j.brs.2011.03.007. Epub 2011 Apr 1. PMID 21777872
- [Background] ter Haar G. Therapeutic applications of ultrasound. Prog Biophys Mol Biol. 2007 Jan-Apr;93(1-3):111-29. doi: 10.1016/j.pbiomolbio.2006.07.005. Epub 2006 Aug 4. PMID 16930682

RESULTS

PARTICIPANT FLOW:
Groups:
- Transcranial Ultrasound: Active stimulation with the transcranial ultrasound at 500 kHz with a duty cycle of 0.24 and pulse repetition frequency of 40 Hz.
  Transcranial Ultrasound: Transcranial ultrasound will be to stimulate at the right fronto-temporal cortex. 30 seconds of stimulation at 500 kHZ with duty cycle 0.24% and pulse rate frequency at 40 Hz.
- Transcranial Ultrasound Sham: Stimulation with the transcranial ultrasound will be on "sham" mode. Unknown to both participants and experimenters, the ultrasound will not stimulate.
  Transcranial Ultrasound: Transcranial ultrasound will be to stimulate at the right fronto-temporal cortex. 30 seconds of stimulation at 500 kHZ with duty cycle 0.24% and pulse rate frequency at 40 Hz.
Period: Overall Study
Arm/Group | Transcranial Ultrasound | Transcranial Ultrasound Sham
Started | 12 | 14
Completed | 12 | 13
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Transcranial Ultrasound | Transcranial Ultrasound Sham | Total
Number analyzed (Participants) | 12 | 14 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 14 | 26
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.58 (.669) | 19.14 (1.292) | 18.88 (1.071)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 18
  Male | 4 | 4 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 3 | 3
  White | 8 | 7 | 15
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 12 | 14 | 26
Beck Depression Inventory II [Mean (Standard Deviation); unit: units on a scale] — The Beck Depression Inventory-II (BDI-II) is one of the most widely used self-report measures for assessing depression. It includes 21 self-report items. Scores range from 0 to 63, and higher scores indicate higher levels of depressive symptoms.
  units on a scale | 17.33 (4.207) | 16.57 (5.36) | 16.92 (4.783)
Penn State Worry Questionnaire [Mean (Standard Deviation); unit: units on a scale] — The PSWQ assesses trait worry, a key component of Generalized Anxiety Disorder. Participants rate themselves on a scale of 1 ("not at all typical of me") to 5 ("very typical of me") for sixteen different statements. Scores range from 16-80, and higher scores reflect higher levels of worry. This scale has been widely used to assess worry and will allow for assessment of worry in the present study (Brown et al., 1992).
  units on a scale | 57.75 (9.555) | 50.71 (10.709) | 53.96 (10.611)
Ruminative Responses Scale [Mean (Standard Deviation); unit: units on a scale] — The Ruminative Responses scale (RRS) consists of 22 statements. It measures rumination, past-focused repetitive thinking that causes and maintains depression. Participants are asked to rate on a scale of 1 (almost never) to 4 (almost always) how much they think about various things (e.g. "think about how alone you feel" and "think about all your shortcomings, failings, faults, mistakes"). Scores range from 22 to 88 with higher scores indicating more rumination.
  units on a scale | 49.92 (8.764) | 43.29 (9.980) | 46.35 (9.847)
Overall Anxiety Severity and Impairment Scale [Mean (Standard Deviation); unit: units on a scale] — The Overall Anxiety Severity and Impairment Scale (OASIS) assesses severity of anxiety symptoms across anxiety disorders and with subsyndromal symptoms. Participants rate five items on a scale from 0 (indicating no anxiety or impairment) to 4 (indicating severe or extreme anxiety or impairment). Scores range from 0 to 20, with higher scores indicating more severe anxiety and impairment from anxiety (Norman et al., 2006).
  units on a scale | 5.75 (3.415) | 5.79 (2.392) | 5.77 (2.847)

OUTCOME MEASURES:

1. Primary Outcome: Depressive Symptoms Assessed With the Beck Depression Inventory-II
Description: The Beck Depression Inventory-II (BDI-II) is one of the most widely used self-report measures for assessing depression. It includes 21 self-report items. Scores range from 0 to 63, and higher scores indicate higher levels of depressive symptoms. In this study, the BDI-II was used to monitor depressive symptoms each day. The outcome is the change in BDI-II score as measured by BDI-II on Day 5 minus BDI-II on Day 1.
Time Frame: Once on day 1 & day 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Transcranial Ultrasound | Transcranial Ultrasound Sham
Number analyzed (Participants) | 12 | 12
units on a scale | -4.42 (4.621) | -.650 (4.249)

2. Secondary Outcome: Rumination Symptoms Assessed With the Ruminative Responses Scale
Description: The Ruminative Responses scale (RRS) consists of 22 statements. It measures rumination, past-focused repetitive thinking that causes and maintains depression. Participants are asked to rate on a scale of 1 (almost never) to 4 (almost always) how much they think about various things (e.g. "think about how alone you feel" and "think about all your shortcomings, failings, faults, mistakes"). Scores range from 22 to 88 with higher scores indicating more rumination. The RRS was used in this study to measure symptoms of rumination on the first and fifth day of this study. The outcome is the difference from Day 5 to Day 1.
Time Frame: Once on day 1 & 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Transcranial Ultrasound | Transcranial Ultrasound Sham
Number analyzed (Participants) | 12 | 12
units on a scale | -1.83 (5.670) | -2.10 (6.045)

3. Secondary Outcome: Worry Symptoms Assessed With the Penn State Worry Questionnaire
Description: The PSWQ assesses trait worry, a key component of Generalized Anxiety Disorder. Participants rate themselves on a scale of 1 ("not at all typical of me") to 5 ("very typical of me") for sixteen different statements. Scores range from 16-80, and higher scores reflect higher levels of worry. This scale has been widely used to assess worry and will allow for assessment of worry in the present study (Brown et al., 1992). The PSWQ was used to monitor symptoms of worry on first and fifth day of this study. The outcome measure is difference from Day 5 to Day 1.
Time Frame: Once on day 1 & day 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Transcranial Ultrasound | Transcranial Ultrasound Sham
Number analyzed (Participants) | 12 | 12
units on a scale | -1.83 (7.732) | 3.30 (5.677)

4. Secondary Outcome: Anxiety Symptoms Assessed With the Overall Anxiety Severity and Impairment Scale
Description: The Overall Anxiety Severity and Impairment Scale (OASIS) assesses severity of anxiety symptoms across anxiety disorders and with subsyndromal symptoms. Participants rate five items on a scale from 0 (indicating no anxiety or impairment) to 4 (indicating severe or extreme anxiety or impairment). Scores range from 0 to 20, with higher scores indicating more severe anxiety and impairment from anxiety (Norman et al., 2006). The OASIS was used to monitor overall severity of anxiety on each day of the study. The outcome measure is difference from Day 5 to Day 1.
Time Frame: Once on day 1 & day 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Transcranial Ultrasound | Transcranial Ultrasound Sham
Number analyzed (Participants) | 12 | 12
units on a scale | -1.33 (1.723) | -2.50 (3.240)

5. Post Hoc Outcome: State Anxiety Assessed With Two Items From the Visual Analogue Mood Scale
Description: The Visual Analog Mood Scale (VAMS) asks patients to rate how much they are experiencing eight mood categories on a scale of 0-100. Global Affect and Global Vigor are subscales. The Global Vigor scale includes a number of items related to anxiety (calm, tense) as well as fatigue (alert, weary). Based on decreases that were seen in global vigor, we create a sum variable of only calm & tense items on the VAMS to examine whether state anxiety decreased. Scores range from 0-20, with higher scores indicating more anxiety. This sum variable served as a post-hoc measures of anxiety each day of the study before stimulation/sham, 10 minutes after stimulation/sham, and 30 minutes after stimulation/sham. Outcome is the difference between measure taken 10 minutes after Stim/Sham and measure taken before Stim/Sham. This measure was taken each of the five days and outcome represents the average over all five days from after to before Stim/Sham.
Time Frame: Assessed before Stim/Sham and 10 minutes after every day for five days; scores represent change from after to before stim/sham averaged across all five days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Transcranial Ultrasound | Transcranial Ultrasound Sham
Number analyzed (Participants) | 12 | 12
units on a scale | -11.9833 (27.24018) | -.6082 (33.90624)

ADVERSE EVENTS:
Time Frame: Participants were monitored for the length of time during which they participated in the study. For most participants, they were monitored from Day 1 of participation to Day 5 of participation (Day 1 to Day 5 occurred within 7 days). However, participants had an option to continue the study up to 10 days if they felt it was helpful for their depression. As such, participants could be monitored for up to 10 days of participation (within 14 days).
Arm/Group | Transcranial Ultrasound | Transcranial Ultrasound Sham
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/14
Other Adverse Events (participants affected / at risk) | 0/12 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes